CLINICAL TRIAL: NCT00629083
Title: A Single-Masked, Randomized, Multi-Center, 2-Arm Parallel Study Comparing the Safety and Effectiveness of Bulkamid® and Contigen® as Bulking Agents for the Treatment of Stress Urinary Incontinence in Females
Brief Title: Bulking Agents for the Treatment of Stress Urinary Incontinence in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contura (Industry)
Collaborators: Regulatory and Clinical Research Institute Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CONSUI-US01
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Results first posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2019-12

CONDITIONS: Stress Urinary Incontinence
Keywords: SUI; Bulkamid; Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 1 (Experimental): Bulkamid Hydrogel injection
  Interventions: Device: Bulkamid
- 2 (Active Comparator): Contigen injection
  Interventions: Device: Contigen

INTERVENTIONS:
Device: Bulkamid — Bulking injection with Bulkamid injection device
  Arms: 1
Device: Contigen — Transurethral bulking injection
  Arms: 2

SUMMARY:
The primary purpose of this study is to demonstrate the safety and effectiveness of Bulkamid® in the treatment of stress urinary incontinence (SUI) due to intrinsic sphincter deficiency (ISD) in adult women who have SUI or stress predominant mixed incontinence

DETAILED DESCRIPTION:
The study is a single-masked, randomized, comparative multi-center, 2-arm parallel study intended to demonstrate the safety and effectiveness of Bulkamid® vs. Contigen® for the treatment of stress urinary incontinence (SUI)due to intrinsic sphincter deficiency (ISD) in adult women who have SUI or stress predominant mixed incontinence.

Subjects will be randomized to receive either a polyacrylamide hydrogel (Bulkamid®) treatment, or a collagen treatment (Contigen®) using a 2:1 ratio and will be masked to the treatment. Screening baseline evaluations and collagen skin testing will be completed to determine eligible subjects. Following a negative skin test, a subject will be randomized and treated with Bulkamid® or the comparator device at the Treatment Visit.

Subjects that are not continent will be considered for re-injection. A maximum of 3 injections (initial + 2 re-injections) are allowed. After the last injection, subjects will attend the 3-Month, 6-Month and 12-Month Follow-up Visits plus a telephone contact at 9 months.

The study will record objective incontinence measurements, subject's perception of effectiveness and quality of life assessments. Adverse events will be recorded throughout the study.

Each subject will be followed for 12 months from the last injection.

ELIGIBILITY:
Inclusion Criteria:

* Be female 18 or more years of age.
* Females of childbearing potential or <2 years post-menopausal must be using 2 forms of contraception.
* Suffer from SUI for at least 6 months.
* Have failed 2 previous non-invasive therapies for 3 months each.
* Have at least 3 incontinence episodes measured over 3 days.
* Have a baseline 24h pad test weight greater than or equal to 5 gm.
* Have VLPP ≤ 100 cm H2O.
* Have maximum cystometric capacity equal or higher than (≥) 250 mL.
* Have PVR urine ≤ 100 mL.
* Have a life expectancy of more than 2 years.

Exclusion Criteria:

* Has urethral hypermobility >30 deg.
* Has predominant urge incontinence.
* Has detrusor overactivity.
* Regularly or intermittently users of urethral catheter.
* Has had previous radiation treatment in the pelvic floor.
* Has had previous urethral surgery (i.e. fistula, diverticula)or urethral bulking. Failed sling or colposuspension procedure for at least 6 months may be included.
* Suffers from known polyuria.
* Has had three (3) or more culture-proven bacterial UTIs in the last 12 months.
* Has a current infection (urethritis, cystitis or vaginitis).
* Has unevaluated hematuria.
* Has a Prolapse Stage greater than II.
* Has a BMI>35 kg/m2.
* Is taking pharmacological treatment for stress urinary incontinence, 4 weeks prior to screening.
* Is allergic to bovine collagen.
* Is known to suffer from severe allergies or anaphylaxis.
* Suffers from autoimmune diseases (e.e. connective tissue diseases) that could confound the treatment.
* Is currently taking or has taken systemic corticosteroids within the past 3 months.
* Currently has cancer or has a history of any cancer within the past 5 years (skin cancer with no evidence of skin malignancy, for at least 2 years, can be included).
* Currently suffering from unstable cardiovascular disease, cancer or uncontrolled diabetes.
* Has active herpes genitalis.
* Is currently participating in any other clinical trial or has participated in another clinical trial within 3 months of screening/baseline visit.
* Is pregnant, lactating or intending to become pregnant.
* Is not physically able to perform study procedure.
* Has a neurogenic bladder
* Had a vaginal delivery within 3 months prior to screening.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Garcia-Codony, Study Director — Contura
Locations (34):
- United States (28):
  - Incontinence Research Institute, Encinitas, California
  - Tower Urology - Institute for Continence - Cedars-Sinai Medical Office, Los Angeles, California
  - Sherif Aboseif, MD, Oxnard, California
  - South California Permanente Medical Group, Pasadena, California
  - Stanford UniveritySchool of Medicine - Departmert of OB/GYN, Stanford, California
  - Genitourinary Surgical Consultants, Denver, Colorado
  - Mayo Clinic - Department of Urology, Jacksonville, Florida
  - University of Miami and Jackson Memorial Hospital, Miami, Florida
  - Specialists in Urology, Naples, Florida
  - Discovery Clinical Trials, Winter Haven, Florida
  - North Shore University Health System, Evanston, Illinois
  - Ochsner Clinic, New Orleans, Louisiana
  - LSU Health Science Center, New Orleans, Louisiana
  - Michigan Urology, Troy, Michigan
  - Northeast Urogynecology, Albany, New York
  - McKay Urology, Charlotte, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - Midwest Institute for Research & Education, West Chester, Ohio
  - St. Lukes Hospital and Health Network, Allentown, Pennsylvania
  - Hospital for the University of Pennsylvannia - Penn Center for Continence and Public Health: Division of Urology, Philadelphia, Pennsylvania
  - Medical University of South Carolina - Department of Urology, Charleston, South Carolina
  - Urology Clinics of North Texas, Dallas, Texas
  - UT Southwestern Medical Center at Dallas - Department of Urology, Dallas, Texas
  - Vanguard Urologic Research Foundation, Houston, Texas
  - Urology San Antonio, San Antonio, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - University of Vermont - The Continence Center, Burlington, Vermont
  - Virgina Mason Medical Center - Section of Urology and Renal Transplantation, Seattle, Washington
- Canada (5):
  - Can-Med Clinical Research, Inc., Victoria, British Columbia
  - Gary Steinhoff Clinical Research, Victoria, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - University of Sherbrooke, Sherbrooke, Quebec
- Hopital Tenon, Paris, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on June 4, 2008, and the last subject was enrolled on June 6, 2011. All participating study centers were in hospitals or clinics in the United States, Canada or France. The sites and investigators were qualified to treat stress urinary incontinence in women by experience and expertise.
Pre-assignment Details: Pelvic Organ Prolapse Quantification, upright cystometry, Valsalva Leak Point Pressure, post-void residual measurement, daily number of incontinence episodes and a 24-hour pad test were completed prior to randomization to confirm eligibility in the trial.
Groups:
- Bulkamid Hydrogel: Bulkamid hydrogel is a proprietary, cross-linked polyacrylamide hydrogel developed for urethral bulking. The hydrogel consists of a backbone of cross-linked polyacrylamide, with water molecules loosely bound to the polymer matrix.
- Contigen Injection: Contigen is a sterile non-pyrogenic implantable device composed of highly purified bovine dermal collagen that was lightly crosslinked with glutaraldehyde and dispersed in phosphate-buffered physiological saline
Period: Overall Study
Arm/Group | Bulkamid Hydrogel | Contigen Injection
Started | 228 | 117
Completed | 200 | 103
Not Completed | 28 | 14
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 3 | 1
Not completed — Withdrawal by Subject | 10 | 2
Not completed — Lost to Follow-up | 12 | 8
Not completed — Moved out of country/state | 2 | 1
Not completed — Refused to return for 12 month visit | 1 | 0

BASELINE CHARACTERISTICS:
Population: There was no difference in the analysis population from the assignment in participant flow.
Groups:
- Bulkamid Hydrogel Injection: Bulkamid: Bulking injection with Bulkamid injection device
- Contigen Injection: Contigen: Transurethral bulking injection
- Total: Total of all reporting groups
Arm/Group | Bulkamid Hydrogel Injection | Contigen Injection | Total
Number analyzed (Participants) | 228 | 117 | 345
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (11.4) | 57.4 (14.3) | 57.8 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 228 | 117 | 345
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 11 | 33
  Not Hispanic or Latino | 206 | 106 | 312
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 214 | 109 | 323
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 31 | 15 | 46
  United States | 197 | 102 | 299
Region of Enrollment [Number; unit: participants]
  Canada | 43 | 21 | 64
  United States | 185 | 96 | 281
24-hour Pad Test [Mean (Standard Deviation); unit: g] — The 24-hour pad test is a standard test used to quantify the amount of urine leaked in a 24-hour period. The patient receives a known quantity and weight of dry pads at a clinic visit, wears them for 24 hours, stores the wet pads in a waterproof/airproof bag, and returns the used and unused pads to the clinic, where they are weighed and the amount of leaked urine (wet pads) is measured by weight. Population: There were 345 subjects enrolled but not all of them provided baseline data for the 24-hour pad test. 223/228 test subjects and 112/117 control subjects provided baseline 24-hour pad test data.
  g
    number analyzed (Participants) | 223 | 112 | 335
    (all) | 93.6 (127.8) | 115.4 (245.9) | 104.5 (186.7)
Daily Number of Incontinence Episodes [Mean (Standard Deviation); unit: number of daily episodes] | 4.1 (2.8) | 3.5 (2.4) | 3.8 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint
Description: The number of subjects with at least a 50% reduction from baseline in both leakage, as measured by the 24h Pad Test, and daily number of incontinence episodes
Time Frame: 12 Months
Population: Intent-to-treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | Bulkamid Hydrogel Injection | Contigen Injection
Number analyzed (Participants) | 228 | 117
participants | 107 | 50

2. Primary Outcome: The Number of Participants With Device- and Procedure-related Serious Adverse Events Through 12 Months Follow-up.
Description: The number of participants with device- and procedure-related serious adverse events through 12 months follow-up.
Time Frame: 12 months
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Bulkamid Hydrogel Injection | Contigen Injection
Number analyzed (Participants) | 228 | 117
Participants | 1 | 0

3. Secondary Outcome: 24hr Pad Test
Description: A measure of urine leaked during a 24-hour period on a known weight and quantity of pads at the 12-month endpoint.
Time Frame: 12 months
Population: Complete Case (CC): Randomized subjects with complete data for a specific endpoint at a particular time point (no imputed data).
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Bulkamid Hydrogel Injection | Contigen Injection
Number analyzed (Participants) | 186 | 94
grams | 32.0 (64.2) | 54.6 (120.3)

4. Secondary Outcome: Number of Subjects Reporting as a Responder
Description: At the 12-month primary endpoint follow-up visit, the subject was asked to provide her perception of treatment effectiveness by circling the most accurate description of her condition: cured/dry; much improved; improved; no change; worse. The response was dichotomized into responder or non-responder. A subject was classified as a responder if she reported that the treatment had cured, much improved, or improved her incontinence condition.
Time Frame: 12 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Bulkamid Hydrogel Injection | Contigen Injection
Number analyzed (Participants) | 187 | 101
Participants | 144 | 71

5. Secondary Outcome: IQoL
Description: The IQoL is a validated instrument consisting of 22 questions grouped into three subscales: avoidance and limiting behaviors; psychosocial impacts, and social embarrassment. It is a subject self-reported quality-of-life measure specific to urinary problems that is used to assess the impact of urinary incontinence and urinary problems and their treatment. The subject scores each question on a scale of 1 to 5 with higher scores indicating more positive responses. The maximum score was 110 points and the minimum score was 22.
Time Frame: 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bulkamid Hydrogel Injection | Contigen Injection
Number analyzed (Participants) | 198 | 103
score on a scale | 80.3 (20.1) | 75.2 (23.3)

6. Secondary Outcome: ICIQ-UI Short Form
Description: The ICIQ-UI Short Form assesses the impact of symptoms of incontinence on quality of life and outcome of treatment. The questionnaire consists of three questions with a maximum score of 21 and a minimum score of zero (0). A lower score represents a decrease in the severity of symptoms (i.e., improvement).
Time Frame: 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bulkamid Hydrogel Injection | Contigen Injection
Number analyzed (Participants) | 196 | 102
score on a scale | 7.1 (4.9) | 7.9 (5.5)

7. Secondary Outcome: Number of Incontinence Episodes
Description: The total number of incontinence episodes experienced by the subject over three consecutive days.
Time Frame: 12 months
Population: This analysis was performed on the Complete Case (CC) analysis set.
Measure: Mean (Standard Deviation); unit: Episodes
Groups:
- Treament: Bulkamid Hydrogel injection
  Bulkamid: Bulking injection with Bulkamid injection device
- Control: Contigen injection
  Contigen: Transurethral bulking injection
Arm/Group | Treament | Control
Number analyzed (Participants) | 195 | 101
Episodes | 1.4 (1.7) | 1.4 (1.9)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from each participant through her study completion visit, typically at 12 months.
Description: The definition of adverse event and/or serious adverse event used to collect adverse event information do not differ from the clinicaltrials.gov definitions.
Arm/Group | Bulkamid Hydrogel Injection | Contigen Injection
All-Cause Mortality (participants affected / at risk) | 0/228 | 0/117
Serious Adverse Events (participants affected / at risk) | 5/228 | 0/117
Other Adverse Events (participants affected / at risk) | 0/228 | 0/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bulkamid Hydrogel Injection (N=228) | Contigen Injection (N=117)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (3) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less